CLINICAL TRIAL: NCT03855410
Title: Preventing Substance Use and HIV/STI Among Urban Youth Via an M-Health Primary Care Preventive Intervention
Brief Title: Preventing Cigarette Use Among Urban Youth Via an M-Health Primary Care Preventive Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David Cordova, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00097290
Record Dates: First submitted 2019-02-15; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Tobacco Use; Drug Use; Adolescent Behavior; Alcohol Use; Sexual Risk Behavior
Keywords: mHealth; preventive intervention; substance use; youth; eHealth; technology-based; HIV/STI
MeSH Terms: conditions — Tobacco Use; Adolescent Behavior; Alcohol Drinking; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: To test the preliminary efficacy of S4E, we will conduct a stage 1 randomized control trial (RCT) and use a mixed between/within-subjects design with two levels of intervention (S4E and Attention-Matched Control) as the between-subjects factor and a repeated measure assessment at 30 days post-Baseline as the within-subject factor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S4E App intervention (Experimental): Participants in the S4E group will receive the tobacco modules via iPads in a private room. The intervention will last approximately 20 minutes. Content includes the theoretically driven components of S4E: (a)Storytelling scenarios, (b) an introduction video, tobacco use knowledge development, (c) interactive activities, (d) increasing self-efficacy to prevent tobacco use, (e) clinician-youth communication, and (f) highlighting prevention principles. Participants in this group also receive usual care. The Clinic's usual care includes a standard risk behaviors intake form, pamphlets highlighting resources on sexual, physical, and mental health, and other healthcare services. Adolescents will be compensated $20 at baseline and $40 at 30-day follow-up. To minimize bias, randomization will occur prior to baseline assessment.
  Interventions: Behavioral: S4E
- Attention-Matched Control (Experimental): Participants in the Attention-Matched Control group will receive a portable document format (PDF) version of the tobacco module content, an enhancement to the care they would receive should they not join the study. Participants in this group also receive usual care. The Clinic's usual care includes a standard risk behaviors intake form, pamphlets highlighting resources on sexual, physical, and mental health, and other healthcare services. Adolescents will be compensated $20 at baseline and $40 at 30-day follow-up. To minimize bias, randomization will occur prior to baseline assessment.
  Interventions: Behavioral: Attention-Matched Control Group

INTERVENTIONS:
Behavioral: S4E — The face-to-face version of S4E (i.e., Storytelling for Empowerment) is registered as a best-practice with the Substance Abuse and Mental Health Services Administration's (SAMHSA) National Registry of Evidence-Based Practices and Programs.The S4E mHealth app was developed in collaboration with youth in Southeast Michigan. Content produced for the application is based on scientific prevention principles in conjunction with youth input. To date, we have developed modules focused on youth alcohol and drug use, HIV and STIs. We now propose to develop modules focused on tobacco prevention and cessation. S4E aims to increase self-efficacy and communication about health risk behaviors. The face-to-face version of S4E has been shown to prevent and reduce substance use, including cigarette use, as well as increase (1) substance use prevention knowledge, (2) communication about health risk behaviors, and (3) perception of harm and self-efficacy in refusing licit and illicit substances.
  Arms: S4E App intervention
Behavioral: Attention-Matched Control Group — Participants in the Attention-Matched Control group will receive a PDF version of the tobacco module material, an enhancement to the usual care they would receive should they not join the study. Participants in this group will also receive usual care. The Clinic's usual care includes standard risk behaviors intake form, pamphlets highlighting resources on sexual, physical, and mental health, and other healthcare services.
  Arms: Attention-Matched Control

SUMMARY:
The study aims to develop tobacco modules to be included in an innovative mobile-health (mHealth) intervention (hereon referred to as S4E) and to determine the feasibility and preliminary efficacy of the updated version of S4E in an urban youth-centered community health clinic in Southeast Michigan.

DETAILED DESCRIPTION:
Tobacco use remains a significant public health concern in the US, and youth are disproportionately affected. Among high school youth , 38% report lifetime cigarette use, and 9.3% report having smoked a whole cigarette before the age of 13. In Southeast Michigan, African-American youth are at disproportionate risk of engaging in tobacco use and co-occuring substance use and other risk behaviors. To address these significant public health concerns, we developed Storytelling 4 Empowerment (S4E), a targeted and tailored mobile-health (mHealth) application (app) intervention to be delivered in health clinic settings. The proposed research aims to develop culturally congruent and developmentally appropriate modules focused on tobacco use prevention and risk reduction to be included as part of the S4E mHealth app. The proposed research will also determine the preliminary efficacy of S4E in reducing tobacco use, alcohol and other drug use, sexual risk behaviors, and improving HIV/STI testing in a sample (n=50) of youth ages 13-21 living in Southeast Michigan.

ELIGIBILITY:
Inclusion Criteria:

* Female, Male, and Transgender adolescents
* Adolescents 13-21 years of age
* Adolescents must live in Southeast Michigan
* Adolescents must provide assent and consent

Exclusion Criteria:

* Report of a prior psychiatric hospitalization by adolescent or caregiver
* Adolescent reports (tentative or firm) plans to move out of the Southeast Michigan area during the study.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Tobacco Use from baseline to 30 days | baseline and 30 days post-baseline
  Tobacco use will be measured at baseline and 30-days post intervention, to assess change in usage.

SECONDARY OUTCOMES:
Change in Drug Use from baseline to 30 days | baseline and 30 days post-baseline
  Licit and illicit drug use behaviors will be assessed using items from the Monitoring the Future study. Youth will be asked whether or not they have used licit or illicit drugs in their lifetime and the past 30 days. Youth who report "YES" to past 30-day drug use will be asked to report the frequency of drug use. These measures have been used in our formative research.
Change in contraception (non-condom) use from baseline to 30 days | baseline and 30 days post-baseline
  Adolescent contraception (non-condom) use will be measured using items extracted from Jemmott, Jemmott, and Fong's Sexual Behavior instrument. This gated instrument will assess the adolescent's past contraceptive use (non-condom) use.
Change in Number of sexual partners from baseline to 30 days | baseline and 30 days post-baseline
  Adolescent number of sexual partners will be measured using items extracted from Jemmott, Jemmott, and Fong's Sexual Behavior instrument. This gated instrument will assess the adolescent's past number of sexual partners.
Change in Alcohol Use from baseline to 30 days | baseline and 30 days post-baseline
  Past 30-day alcohol use behaviors will be assessed using items from the Monitoring the Future study. Youth will be asked whether or not they have used alcohol in their lifetime and the past 30 days. Youth who report "YES" to past 30-day alcohol use will be asked to report the frequency of alcohol use. These measures have been used in our formative research.
Change in Binge Drinking from baseline to 30 days | baseline and 30 days post-baseline
  Past 2-weeks binge drinking behaviors will be assessed using items from the Monitoring the Future study. Youth will be asked whether or not they have had 5 or more drinks of alcohol in a row within a couple of hours in the past 2-weeks. Youth who report "YES" to past binge drinking will be asked to report the frequency of binge drinking. These measures have been used in our formative research.
Change in Unprotected sex from baseline to 30 days | baseline and 30 days post-baseline
  Condom use behaviors will be assessed. Youth will be asked whether they are sexually active or not. Youth who report "YES" to being sexually active will be asked to report whether or not they have had unprotected sex in their lifetime and past 30-days and the frequency of unprotected sex, if they used condoms the last time they had sex, and if they plan on using condoms next time. These measures have been used in our formative research.
Change in alcohol or drug use before sex from baseline to 30 days | baseline and 30 days post-baseline
  Alcohol or drug use before sex will be assessed. Youth will be asked whether they have used alcohol or drugs before sex in their lifetime and past-30 days. Youth who report "YES" will be asked to report the frequency of alcohol and drug use before sex. These measures have been used in our formative research.
Change in HIV/STI testing from baseline to immediately post-intervention and 30 day post-intervention | baseline, immediately post-intervention, and 30 days post-intervention
  HIV/STI testing will be assessed. Youth will be asked to report lifetime HIV and STI testing, whether or not they received an HIV or STI test during the clinic visit, and HIV or STI testing in the past 30-days. Additionally, clinicians will be asked whether or not their youth participant received an HIV or STI test during the clinic visit. These measures have been used in our formative research

OTHER OUTCOMES:
Change in Clinician-Youth Communication for Clinicians from baseline to immediately post-intervention and 30 days post-intervention | baseline, immediately post-intervention, and 30 days-post baseline
  Completed by the clinician, clinician-youth communication will be assessed post-baseline using items adapted from the Matched Pair Instrument (19 items; MPI). MPI assesses process and content of communication, including verbal and action-related behaviors performed by clinicians. Responses range from "1=strongly disagree," to "5=strongly agree," on a five-point Likert scale. A sample statement for clinicians and youths is, "I encouraged the patient to express his or her thoughts concerning drug use behaviors."
Change in Clinician-Youth Communication for Youth from baseline to immediately post-intervention and 30 days post-intervention | baseline, immediately post-intervention, and 30 days-post baseline
  Completed by the youth, clinician-youth communication will be assessed post-baseline using items adapted from the Matched Pair Instrument (19 items; MPI). MPI assesses process and content of communication, including verbal and action-related behaviors performed by clinicians. Responses range from "1=strongly disagree," to "5=strongly agree," on a five-point Likert scale. A sample statement for youths is, "I was encouraged to express my thoughts concerning drug use behaviors."
Change in Youth Self-Efficacy as measured by the Condom Self-Efficacy Scale from baseline to immediately post-intervention and 30 days post-intervention | baseline, immediately post-intervention, and 30 days-post baseline
  Youth's self-efficacy will be assessed using the Condom Self-Efficacy Scale (19 items, α =.85). Responses range from "1=not sure at all," to "4=definitely sure," on a four-point Likert scale. A sample question for the youth is, "How sure are you that you can refuse if a friend offers you marijuana at a party and you do not want it?"
Change in Youth Self-Efficacy as measured by Drug Use Resistance Self-Efficacy Scale from baseline to immediately post-intervention and 30 days post-intervention | baseline, immediately post-intervention, and 30 days-post baseline
  Youth's self-efficacy will be assessed using the Drug Use Resistance Self-Efficacy (24 items, α =.98). Responses range from "1=not sure at all," to "4=definitely sure," on a four-point Likert scale. A sample question for the youth is, "How sure are you that you can refuse if a friend offers you marijuana at a party and you do not want it?"

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Corner Health Center, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordova D, Alers-Rojas F, Lua FM, Bauermeister J, Nurenberg R, Ovadje L, Fessler K, Delva J, Salas-Wright CP, Council YL. The Usability and Acceptability of an Adolescent mHealth HIV/STI and Drug Abuse Preventive Intervention in Primary Care. Behav Med. 2018 Jan-Mar;44(1):36-47. doi: 10.1080/08964289.2016.1189396. Epub 2016 Jul 15. PMID 27223646
- [Background] Cordova D, Bauermeister JA, Fessler K, Delva J, Nelson A, Nurenberg R, Mendoza Lua F, Alers-Rojas F, Salas-Wright CP; Youth Leadership Council. A Community-Engaged Approach to Developing an mHealth HIV/STI and Drug Abuse Preventive Intervention for Primary Care: A Qualitative Study. JMIR Mhealth Uhealth. 2015 Dec 18;3(4):e106. doi: 10.2196/mhealth.4620. PMID 26685288
- [Background] Cordova D, Lua FM, Ovadje L, Fessler K, Bauermeister JA, Salas-Wright CP, Vaughn MG, Leadership Council Y. Adolescent Experiences of Clinician-Patient HIV/STI Communication in Primary Care. Health Commun. 2018 Sep;33(9):1177-1183. doi: 10.1080/10410236.2017.1339379. Epub 2017 Jul 7. PMID 28686489
- [Derived] Cordova D, Munoz-Velazquez J, Mendoza Lua F, Fessler K, Warner S, Delva J, Adelman N; Youth Leadership Council; Fernandez A, Bauermeister J. Pilot Study of a Multilevel Mobile Health App for Substance Use, Sexual Risk Behaviors, and Testing for Sexually Transmitted Infections and HIV Among Youth: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Mar 17;8(3):e16251. doi: 10.2196/16251. PMID 32181747